CLINICAL TRIAL: NCT05576428
Title: Efficacy of N-Acetylcysteine in Improving/Normalizing ALT & AST in Patients of NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tazeen Rasheed, Associate Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAFLD-NAC
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DIET& EXERCISE (Active Comparator): diet plan & daily 20 minutes brisk walking.
  Interventions: Behavioral: Diet and exercise
- N Acetylcysteine WITH DIET & EXERCISE (Experimental): NAC 200mg BD along with diet plan & exercise.
  Interventions: Behavioral: Diet and exercise; Drug: NAC with diet and exercise

INTERVENTIONS:
Behavioral: Diet and exercise — diet and exercise in patients of NAFLD
Drug: NAC with diet and exercise — NAC with diet and exercise in patients of NAFLD
  Arms: N Acetylcysteine WITH DIET & EXERCISE

SUMMARY:
Currently researches are focusing on the effect of antioxidants in the treatment of non-alcoholic fatty liver disease (NAFLD). Since N-acetyl cysteine (NAC) has been proven to have antioxidant and anti-inflammatory properties, therefore, we will conduct this study to determine the effect of NAC in patients of NAFLD with raised liver enzymes.

DETAILED DESCRIPTION:
The prevalence of non-alcoholic fatty liver disease (NAFLD) is increasing globally, and presents a challenge for the medical community since it has no FDA approved treatment. An important feature of non-alcoholic fatty liver disease (NAFLD) is hepatic steatosis leading to hepatic dysfunction . It has been reported that NAFLD patients with increased liver enzymes have a greater risk of developing complications like cirrhosis and end-stage liver disease. since N-acetyl cysteine (NAC) has been proven to have antioxidant and anti-inflammatory properties, therefore, we will conduct this study to determine the effect of NAC in patients of NAFLD with raised liver enzymes (ALT, AST). Patients presenting with ultrasound showing fatty liver with raised liver enzymes will be recruited. They will be randomized into two groups (group A and group B).

The odd number patients will be allocated group A and even number patients will be allocated to group B.

Group A: patients in this group will be advised to follow a diet plan & daily 20 minutes brisk walking.

Group B: Patients in this group will be given NAC 200mg BD along with diet plan & exercise. This drug will be provided to the patients by the investigators free of cost.

The liver function tests and side effects of NAC will be followed at 12 weeks .

ELIGIBILITY:
Inclusion Criteria:

* • Patients of both genders between the ages of 20 years and 60 years, giving consent to be included in the study.

  * Patients having fatty liver on ultrasound with raised ALT and AST levels

Exclusion Criteria:

* • Patients having other causes of steatosis eg, excessive alcohol consumption,

  * Patients taking steatogenic medications such as, methotrexate , corticosteroids etc.
  * Patients suffering from other diseases that could increase ALT levels eg. Viral hepatitis, HIV, autoimmune liver diseases, infiltrative liver diseases.
  * Patients suffering from malignancies.
  * Patients who are not compliant to the medicine.
  * Pregnant and nursing females

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in Alanine transaminase,aspartate aminotransferase | 12 weeks
  Change in Alanine transaminase,aspartate aminotransferase

SECONDARY OUTCOMES:
Side Effects of NAC | 12 weeks
  Side Effects of NAC

IPD SHARING:
Plan to Share IPD: No